CLINICAL TRIAL: NCT03575767
Title: Characteristics and Dynamics of TCR Repertoire in Peripheral Blood of Patients With Hematological Malignancies After Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Characteristics and Dynamics of TCR Repertoire in Patients With Hematological Malignancies After Allo-HSCT
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Hangzhou ImmuQuad Biotechnologies, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 307-TCR-NGS-001
Record Dates: First submitted 2018-06-21; First posted 2018-07-03 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Hematologic Neoplasms; Hematopoietic Stem Cell Transplantation; Graft Vs Host Disease; Recurrence
Keywords: TCR Repertoire; Next Generation Sequencing; ALL; AML; MDS; Myeloablative
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Myeloablative Hematopoietic Stem Cell Transplantation — Myeloablative hematopoietic stem cell transplantation from many kinds of donors, including matched related donor, matched unrelated donor, haploidentical related donor.

SUMMARY:
Graft-versus-Host Disease (GVHD) and relapse, which is mainly due to lack of Graft-versus-Leukemia (GVL), are the most frequent and severe complications of allogeneic hematopoietic stem cell transplantation (allo-HSCT). T cells expanded from mature T cells in the graft play a dominant role in development of GVHD and GVL early after allo-HSCT. Recent applications of high-throughput sequencing (HTS) to the T cells repertoire open a new avenue for us to look deeply into how these T cells dynamically adjust in the context of the recipient's environment.

The main goal of this research study is to set up a mathematical model based on T cell receptor (TCR) sequencing to enable prediction for the key immunologic outcomes early post-transplantation. This study will deepen the understanding of the molecular mechanisms driving the most deadly post-transplantation complications, and serve as convincing evidence upon which to choose a better donor and a more proper transplantation approach.

This observational trial will perform HTS for TCR β-chain complementarity determining region 3 (CDR3) repertoires of grafts and peripheral blood samples from recipients post-transplantation and analyze the relationship between dynamics of TCR CDR3 repertoires and clinical outcomes early post-transplantation, especially including GVHD and relapse. The investigators want to know how the antigen environment in recipients drives dynamics of mature T cells from grafts in order to use the new discovered rules to better predict and treat the disease process.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AML, ALL, MDS, undergone myeloablative hematopoietic stem cell transplantation about 1 year ago.
2. Patients who have residual peripheral blood mononuclear cell samples freezed up to now which had been disposed at the time of about 1-month, 2-month after allo-HSCT.
3. Patients whose residual grafts have been freezed up to now.

Exclusion Criteria:

1. Patients whose grafts or residual peripheral blood mononuclear cell samples are failed to be thawed.
2. Patients whose samples are failed with RNA extraction.
3. Patients whose RNA sequencing are failed.
4. Patients who died within 2 months after allo-HSCT.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients undergone myeloablative hematopoietic stem cell transplantation about 1 year ago.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Perform TCR β-chain CDR3 high-throughput sequencing and TCR repertoire analysis on T cells from the graft and the peripheral blood at the time of 1-month, 2-month after allo-HSCT. | 3 months
  To identify the mechanisms specific for TCR repertoire dynamics and rearrangement characteristics.

SECONDARY OUTCOMES:
Perform longitudinal immune analysis on T cells purified from patients undergoing allogeneic HSCT who develop acute and chronic GVHD, relapse, and virus infectious complications post-transplant. | 1 year
  Characterize the main TCR β-chain CDR3 sequences dynamic change responsible for acute GVHD, chronic GVHD and defects in protective immunity in patients undergoing HSCT.
Perform horizontal comparison analysis on the diversity index of T cells purified from the grafts and the patients undergoing allogeneic HSCT. | 1 year
  Characterize the TCR β-chain CDR3 repertoire dynamic change responsible for acute GVHD, chronic GVHD and defects in protective immunity in patients undergoing HSCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, Beijing Municipality, China